CLINICAL TRIAL: NCT04948762
Title: A Contemporary Review of Surgical Approaches in Pelvic Exenterative Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Des Winter, Professor Desmond C Winter, St Vincent's University Hospital, Ireland
Other Study IDs: PelvEx 5
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Pelvic Exenteration; Advanced Pelvic Malignancy; Locally Advanced Rectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open: Patients who underwent an open approach to pelvic exenteration
- Laparoscopic: Patients who underwent a laparoscopic approach to pelvic exenteration
- Robotic: Patients who underwent a robotically-assisted pelvic exenteration

SUMMARY:
Minimally-invasive surgery (MIS) techniques have revolutionised the approach to rectal cancer surgery. With increasing experience, surgeons have began to utilise these platforms increasingly in the context of pelvic exenteration (PE). This observational retrospective review plans to assess the volume of PE being performed on a global basis and to assess the comparative outcomes associated with each technique in order to assess the optimal approach to radical pelvic surgery.

DETAILED DESCRIPTION:
Pelvic exenteration (extended pelvic multi-visceral resection) is a radical procedure that offers potential long-term cure in appropriately selected cases of locally advanced and recurrent pelvic cancers. It was first described by Alexander Brunschwig in 1948 as a viable palliative option for advanced gynaecological cancer. However, over the last 70 years, changes in surgical oncology practices have seen its role extended to include other advanced non-gynaecological cancers (locally advanced colorectal, urological, and sarcomatous neoplasms).

Although these procedures pose a significant challenge for the operating surgeon, improved surgical techniques, technology, and reconstructive options have facilitated more radical resections. Despite improved surgical options, patients still have considerable post-operative morbidity and negative impact to quality of life. However, non-surgical management options result in poor prognosis with only 3% survival at five-years. Pelvic exenteration in appropriately-selected patients offers the only hope of long-term survival.

Over the last few decades with improved perioperative management and better surgical techniques, more aggressive visceral, soft tissue and bony resections are performed. The development of minimally invasive surgery (MIS) platforms has also evolved substantially, especially regarding pelvic surgery. There are some recent sporadic (low-volume) reports highlighting the potential role for MIS exenterative surgery, however many reports have been heterogeneous and single-centre. The aim of this retrospective review is to compare the volume, disease characteristics and surgical outcomes between open, laparoscopic and robotic pelvic exenterations, and to assess the initial experience of MIS platforms in multiple specialist centres worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or recurrent RECTAL cancer
* Aged over 18 years
* Undergoing a multi-visceral extended pelvic resection
* Procedure took place within the specified timeframe (July 2016 - July 2021)

Exclusion Criteria:

* Extra-pelvic/ non-resectable metastatic or peritoneal disease
* Palliative pelvic exenteration
* Insufficient patient follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are undergoing surgery for histologically-confirmed locally advanced or recurrent rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Resection status | July 2016 - July 2021
  Completeness of the surgical resection (R0, R1 or R2)

SECONDARY OUTCOMES:
Blood loss | July 2016 - July 2021
  Blood loss (mL)
Operation time | July 2016 - July 2021
  Time from first incision to skin closure (minutes)
Conversion rate | July 2016 - July 2021
  Need to convert from robotic or laparoscopic to open procedure
Morbidity | July 2016 - July 2021
  Frequency of post-operative complication, as measured by the Clavien-Dindo scale
Length of stay | July 2016 - July 2021
  Duration of stay in hospital post-procedure
Analgesic Requirements | July 2016 - July 2021
  Quantity of analgesia consumed, primarily opioid analgesia measured in morphine equivalents
Return of bowel function | July 2016 - July 2021
  Time to passage of flatus or bowel motion

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Winter, MD, Study Chair — St. Vincent's Healthcare Group
Locations (1):
- St. Vincent's Hospital, Dublin, Ireland